CLINICAL TRIAL: NCT02229955
Title: A Multicenter, Randomized, Double-blind Phase Ⅲ Study of Cyclosporine Ophthalmic Soution Group and Cyclosporine Ophthalmic Suspension Group 12 Weeks After Treatment in Moderate to Severe Dry Eye Disease
Brief Title: Study of Tisporin Eye Drops Group and Restasis Eye Drops Group After Treatment, Each Treatment Group Comparisons for Evaluation of Efficacy and Safety in Moderate to Severe Dry Eye Disease
Acronym: HL_TSPR_302
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HL_TSPR_302
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Dry Eye Syndromes
Keywords: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- T-sporin eye drop (Experimental): Cyclosporine 0.05% : 1 drop twice a day for 12 weeks to both eyes
  Interventions: Drug: Cyclosporine ophthalmic solution
- Restasis eye drop (Active Comparator): Cyclosporine 0.05% : 1 drop twice a day for 12 weeks to both eyes
  Interventions: Drug: Cyclosporine ophthalmic solution

INTERVENTIONS:
Drug: Cyclosporine ophthalmic solution — 1 drop twice/day for 12 weeks to both eyes
  Other Names: Restasis Eye Drops; Tisporin Eye Drops

SUMMARY:
The purpose of this clinical Study is Tisporin Eye Drops 0.05%(Cyclosporine ophthalmic solution) group and Restasis Eye Drops 0.05%(Cyclosporine ophthalmic suspension) group 12 weeks after treatment, each treatment group comparisons for evaluation of efficacy and safety in Moderate to Severe Dry Eye Disease.

- Corneal staining test, Ocular surface disease index (OSDI), Tear break up time (TBUT), Non-anesthetic Schirmer test

ELIGIBILITY:
Inclusion Criteria:

[Patients with moderate-to-severe ocular dry eye]

1. The One eye of corneal fluorescein staining score of 2 or higher (Oxford grading)
2. Non-anesthetic Schirmer test value ≤ 10mm/5min patients at least one eye score (Non-anesthetic Schirmer test value = 0/5min, nasal stimulation in the same eye, Schirmer test value ≥ 3mm/5min)
3. Tear break-up time is 10 seconds or less
4. Screening both eyes, the corrected visual acuity is 0.2 or more
5. Despite conventional treatment, the symptoms of dry eye signs (Artificial tear eye drops, sympathetic nervous system stimulant agent, parasympathetic nerve stimulant, etc.)

Exclusion Criteria:

1. Screening visits in the previous 3 months (12 weeks) who participated in the clinical trials of cyclosporine eye drops, or if you used a cyclosporin ophthalmic solutions.
2. The patients with systemic or ocular disorders affected the test results (ocular surgery, trauma, or disease)

   1. Abnormal eyelid function : Disoders of the eyelids or eyelashes
   2. Ocular allergies or currently under the treatment of allergic diseases of the eye (topical ocular mast cell stabilizer, antihistamine use, etc.)
   3. Cicatricial keratoconjunctivitis caused by herpetic keratopathy, conjunctival scarring (alkali damage, Steven-Johnson syndrome, cicatricial pemphigoid), pterygium, pinguecula, lack of congenital lacrimal, neurogenic keratitis, keratoconus, corneal transplantation
3. current or recent patients used dry eye syndrome medications (topical or systemic) that may affect the status
4. The use in clinical trials of drug hypersensitivity reactions in patients

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Corneal staining test | 12 weeks

SECONDARY OUTCOMES:
Corneal staining test | 4, 8 weeks
Ocular surface disease index (OSDI) | 4, 8, 12 weeks
Tear break up time (TBUT) | 4, 8, 12 weeks
Non-anesthetic Schirmer test | 4, 8, 12 weeks
Conjunctival staining | 4, 8, 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The catholic university of Korea seoul st. Mary's hospital, Seoul, Seocho-Ku, South Korea